CLINICAL TRIAL: NCT02966574
Title: Magnetic Resonance Imaging of the Whole Body, Including Diffusion, in the Medical Evaluation of Breast Cancers at High Risk for Metastasis and the Follow-up of Metastatic Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Mieke Cannie, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-IRM CE
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breastcancer
Keywords: Whole body MRI; Breastcancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metastatic breast cancer (Experimental)
  Interventions: Device: whole body MRI

INTERVENTIONS:
Device: whole body MRI — The examination will be conducted in the pretreatment assessment of breast cancers with a high metastasis risk and in the monitoring of metastatic breast cancers. The examination is performed without intravenous injection of contrast medium, from the top of the skull to mid-thigh using diffusion weighted sequences in the axial plane, T1-weighted sequences in the coronal plane, STIR T2 weighted sequences in the coronal plane and T1-weighted sequences in the sagittal plane on the spine. Total examination duration is one hour. The interpretation of the results is made by two independent reporters with a complementary expertise, according to a systematic lecture grid.

SUMMARY:
Whole-body MRI including diffusion is a booming technique. Numerous studies have demonstrated its interest in metastatic cancers. Breast cancers, especially hormone-sensitive ones, are very osteophilic and bones are the most frequent metastatic site.

Apart from morphological criteria (lesion size and RECIST criteria), MRI provides quantitative functional criteria (diffusion and ADC values). According to a recent study, whole body MRI is as good as PET/CT and more effective than bone scintigraphy for the diagnosis of bone metastases for cancers of breast and prostate with a high metastatic risk.

Therefore, it seems appropriate to study the performance of whole body MRI in the pre-therapeutic assessment of breast cancer with a high risk for metastasis and the monitoring of metastatic breast cancer.

DETAILED DESCRIPTION:
Whole-body MRI including diffusion is a booming technique. Numerous studies have demonstrated its interest in metastatic cancers.

Breast cancers, especially hormone-sensitive ones, are very osteophilic and bones are the most frequent metastatic site. Other sites include the lungs, liver, pleura, distant lymph nodes, soft tissue and the central nervous system.

Metastasis are located exclusively in the bones in 30% of the cases. The most commonly affected bones include the axial skeleton, rich in hematopoietic bone marrow : column, pelvis, skull, ribs, clavicles, the proximal part of the femur and humerus. Five percent of breast cancers are directly metastatic and 20 to 30% of localized breast cancers progress to metastatic stage. This potentially affects a large number of patients, with a median survival of 30 to 36 months.Patients with bone metastases only have a better survival rate than others: 20% at 5 years. It is therefore important to use a reliable and reproducible examination for the monitoring of treatment response.

Apart from morphological criteria (lesion size and RECIST criteria), MRI provides quantitative functional criteria (diffusion and ADC values). According to a recent study, whole body MRI is as good as PET/CT and more effective than bone scintigraphy for the diagnosis of bone metastases for cancers of breast and prostate with a high metastatic risk. However, this is a preliminary study with a limited and heterogeneous cohort of patients.

Therefore, it seems appropriate to study the performance of whole body MRI in the pre-therapeutic assessment of breast cancer with a high risk for metastasis and the monitoring of metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast carcinoma B5
* Axillary lymph node punction C5 or metastatic
* Performance status from 0 to 2.

Exclusion Criteria:

* Ferromagnetic metallic foreign bodies (pacemakers, implanted cochlear, neurostimulator, ...)
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Apparent diffusion coefficient (ADC) (mm2/sec) | Once per year for a maximum of 2 years
  Apparent diffusion coefficient (ADC) expressed in mm2/sec. Magnetic resonance images realised with the Ingenia 3 Tesla Engine (Philips) and the Area 1,5 Tesla Engine (Siemens).Post-processing realized with the Syngo Onco Care application of Siemens.
Number of cancer lesions | Once per year for a maximum of 2 years
Exact localisation of cancer lesions | Once per year for a maximum of 2 years
  Systematic lecture grid. Possible choices are:
  Nodes (Axillary, internal mammary, supra and infraclavicular, cervical, mediastinal, hilar, upper abdomen, pelvic, inguinal), Bone (Spine, Scapular Belt, Costal Grill, Pelvic Belt)- Lungs and pleura - Liver (and other viscera)- Soft tissues and skin- Brain and spinal cord- Other

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Hottat, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bidard FC, Vincent-Salomon A, Gomme S, Nos C, de Rycke Y, Thiery JP, Sigal-Zafrani B, Mignot L, Sastre-Garau X, Pierga JY; Institut Curie Breast Cancer Study Group. Disseminated tumor cells of breast cancer patients: a strong prognostic factor for distant and local relapse. Clin Cancer Res. 2008 Jun 1;14(11):3306-11. doi: 10.1158/1078-0432.CCR-07-4749. PMID 18519757
- [Background] Senkus E, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rutgers E, Zackrisson S, Cardoso F; ESMO Guidelines Committee. Primary breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v8-30. doi: 10.1093/annonc/mdv298. No abstract available. PMID 26314782
- [Background] Pasoglou V, Michoux N, Peeters F, Larbi A, Tombal B, Selleslagh T, Omoumi P, Vande Berg BC, Lecouvet FE. Whole-body 3D T1-weighted MR imaging in patients with prostate cancer: feasibility and evaluation in screening for metastatic disease. Radiology. 2015 Apr;275(1):155-66. doi: 10.1148/radiol.14141242. Epub 2014 Dec 15. PMID 25513855
- [Background] Dimopoulos MA, Hillengass J, Usmani S, Zamagni E, Lentzsch S, Davies FE, Raje N, Sezer O, Zweegman S, Shah J, Badros A, Shimizu K, Moreau P, Chim CS, Lahuerta JJ, Hou J, Jurczyszyn A, Goldschmidt H, Sonneveld P, Palumbo A, Ludwig H, Cavo M, Barlogie B, Anderson K, Roodman GD, Rajkumar SV, Durie BG, Terpos E. Role of magnetic resonance imaging in the management of patients with multiple myeloma: a consensus statement. J Clin Oncol. 2015 Feb 20;33(6):657-64. doi: 10.1200/JCO.2014.57.9961. Epub 2015 Jan 20. PMID 25605835
- [Background] Woolf DK, Padhani AR, Makris A. Assessing response to treatment of bone metastases from breast cancer: what should be the standard of care? Ann Oncol. 2015 Jun;26(6):1048-1057. doi: 10.1093/annonc/mdu558. Epub 2014 Dec 3. PMID 25471332
- [Background] Jambor I, Kuisma A, Ramadan S, Huovinen R, Sandell M, Kajander S, Kemppainen J, Kauppila E, Auren J, Merisaari H, Saunavaara J, Noponen T, Minn H, Aronen HJ, Seppanen M. Prospective evaluation of planar bone scintigraphy, SPECT, SPECT/CT, 18F-NaF PET/CT and whole body 1.5T MRI, including DWI, for the detection of bone metastases in high risk breast and prostate cancer patients: SKELETA clinical trial. Acta Oncol. 2016;55(1):59-67. doi: 10.3109/0284186X.2015.1027411. Epub 2015 Apr 2. PMID 25833330